CLINICAL TRIAL: NCT06099366
Title: Treatment of Newly Diagnosed Standard Risk Acute Lymphoblastic Leukemia in
Brief Title: Treatment of Newly Diagnosed Standard Risk Acute Lymphoblastic Leukemia in Children
Acronym: SR ALL
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hee Young Ju (Other)
Collaborators: Asan Medical Center (Other); Seoul National University Hospital (Other); Seoul St. Mary's Hospital (Other); Severance Hospital (Other); Pusan National University Yangsan Hospital (Other); Korea University Anam Hospital (Other); Chonnam National University Hospital (Other); Jeju National University Hospital (Other)
Responsible Party: Sponsor-Investigator, Hee Young Ju, Clinical Professor, Samsung Medical Center
Organization: Samsung Medical Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-09-142
Record Dates: First submitted 2023-10-18; First posted 2023-10-25 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Lymphoblastic Leukemia in Children
Keywords: Standard Risk ALL; NGS MRD
MeSH Terms: interventions — Asparaginase; Dexamethasone; Cyclophosphamide; Cytarabine; Methotrexate; Mercaptopurine; Doxorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Standard-low (SL) (Experimental): Induction-> SL Consolidation(4weeks)-> Interim Maintenance 1st-> Delayed Intesificaion-> Interim Maintenance 2nd-> Maintenance
  Interventions: Drug: induction: vincristine, L-asparaginase, dexamethasone, intrathecal Ara-C, intrathecal Methotrexate; Drug: Consolidation: Vincristine, Mecaptopurine, Intrathecal Methotrexate; Drug: Interim Maintenance(IM): Vincristine, Methotrexate, Intrathecal Methotrexate; Drug: Delayed Intesification(DI): Vincristine, Mercaptopurine, L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Dexamethasone, Intrathecal Methotrexate; Drug: Maintenance: Vincristine, Mercaptopurine, Methotrexate, Dexamethasone, Intrathecal Methotrexate
- Standard-average (SA) (Experimental): Induction-> SH Consolidation(4weeks)-> Intensified Consolidation(4weeks)-> Interim Maintenance 1st-> Delayed Intesificaion-> Interim Maintenance 2nd-> Maintenance
  Interventions: Drug: induction: vincristine, L-asparaginase, dexamethasone, intrathecal Ara-C, intrathecal Methotrexate; Drug: Consolidation: Vincristine, Mecaptopurine, Cyclophosphamide, Cytarabine, L-asparaginase, Intrathecal Methotrexate; Drug: Interim Maintenance(IM): Vincristine, Methotrexate, Intrathecal Methotrexate; Drug: Delayed Intesification(DI): Vincristine, Mercaptopurine, L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Dexamethasone, Intrathecal Methotrexate; Drug: Maintenance: Vincristine, Mercaptopurine, Methotrexate, Dexamethasone, Intrathecal Methotrexate
- Standard-high 1 (SH1) (Experimental): Induction-> SL Consolidation(4weeks)-> Intesified Consolidattion(4weeks)-> Interim Maintenance 1st-> Delayed Intesificaion 1st-> Interim Maintenance 2nd-> Delayed Intestificaion 2nd-> Maintenance
  Interventions: Drug: induction: vincristine, L-asparaginase, dexamethasone, intrathecal Ara-C, intrathecal Methotrexate; Drug: Consolidation: Vincristine, Mecaptopurine, Cyclophosphamide, Cytarabine, L-asparaginase, Intrathecal Methotrexate; Drug: Interim Maintenance(IM): Vincristine, Methotrexate, Mercaptopurine, Intrathecal Methotrexate; Drug: Delayed Intesification(DI): Vincristine, L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Dexamethasone, Intrathecal Methotrexate; Drug: Maintenance: Vincristine, Mercaptopurine, Methotrexate, Dexamethasone, Intrathecal Methotrexate
- Standard-high 2 (SH2) (Experimental): Induction-> SH Consolidation(4weeks)-> Intensified Consolidation(4weeks)-> Interim Maintenance 1st-> Delayed Intesificaion 1st-> Interim Maintenance 2nd-> Delayed Intestificaion 2nd-> Maintenance
  Interventions: Drug: induction: vincristine, L-asparaginase, dexamethasone, intrathecal Ara-C, intrathecal Methotrexate; Drug: Consolidation: Vincristine, Mecaptopurine, Cyclophosphamide, Cytarabine, L-asparaginase, Intrathecal Methotrexate; Drug: Interim Maintenance(IM): Vincristine, Methotrexate, Mercaptopurine, Intrathecal Methotrexate; Drug: Delayed Intesification(DI): Vincristine, L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Dexamethasone, Intrathecal Methotrexate; Drug: Maintenance: Vincristine, Mercaptopurine, Methotrexate, Dexamethasone, Intrathecal Methotrexate

INTERVENTIONS:
Drug: induction: vincristine, L-asparaginase, dexamethasone, intrathecal Ara-C, intrathecal Methotrexate — vincristine 1.5mg/m2 L-asparaginase 6,000U/m2 Dexamethasone 6mg/m2 Intrathecal Cytarabine Intrathecal Methotreate
Drug: Consolidation: Vincristine, Mecaptopurine, Intrathecal Methotrexate — Vincristine 1.5mg/m2 Mecaptopurine 50mg/m2 Cyclophosphamide 1,000mg/m2 Cytarabine 75mg/m2 L-asparaginase 6,000U/m2 Intrathecal Methotrexate
  Arms: Standard-low (SL)
Drug: Consolidation: Vincristine, Mecaptopurine, Cyclophosphamide, Cytarabine, L-asparaginase, Intrathecal Methotrexate — Vincristine 1.5mg/m2 Mecaptopurine 50mg/m2 Cyclophosphamide 1,000mg/m2 Cytarabine 75mg/m2 L-asparaginase 6,000IU/m2 Intrathecal Methotrexate
  Arms: Standard-average (SA); Standard-high 1 (SH1); Standard-high 2 (SH2)
Drug: Interim Maintenance(IM): Vincristine, Methotrexate, Intrathecal Methotrexate — Vincristine 1.5mg/m2 Methotrexate 5,000mg/m2 Intrathecal Methotrexate
  Arms: Standard-average (SA); Standard-low (SL)
Drug: Interim Maintenance(IM): Vincristine, Methotrexate, Mercaptopurine, Intrathecal Methotrexate — Vincristine 1.5mg/m2 Methotrexate 5,000mg/m2 Mecaptopurine: 25mg/m2 Intrathecal Methotrexate
  Arms: Standard-high 1 (SH1); Standard-high 2 (SH2)
Drug: Delayed Intesification(DI): Vincristine, Mercaptopurine, L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Dexamethasone, Intrathecal Methotrexate — Vincristine 1.5mg/m2 Mercaptopurine 50mg/m2 L-asparaginase 6,000IU/m2 Doxorubicin 25mg/m2 Cyclophosphamide 1,000mg/m2 Cytarabine 75mg/m2 Dexamethasone 10mg/m2 Intrathecal Methotrexate
  Arms: Standard-average (SA); Standard-low (SL)
Drug: Delayed Intesification(DI): Vincristine, L-asparaginase, Doxorubicin, Cyclophosphamide, Cytarabine, Dexamethasone, Intrathecal Methotrexate — Vincristine 1.5mg/m2 L-asparaginase 6,000IU/m2 Doxorubicin 25mg/m2 Cyclophosphamide 1,000mg/m2 Cytarabine 100mg/m2 Dexamethasone 6mg/m2 Intrathecal Methotrexate
  Arms: Standard-high 1 (SH1); Standard-high 2 (SH2)
Drug: Maintenance: Vincristine, Mercaptopurine, Methotrexate, Dexamethasone, Intrathecal Methotrexate — Vincristine 1.5mg/m2 Mercaptopurine 50mg/m2 Methotrexate 20mg/m2 Dexamethasone 6mg/m2 Intrathecal Methotrexate

SUMMARY:
Aim of this study is to investigate the outcome of NGS MRD based risk stratified treatment for high risk acute lymphoblastic leukemia in children and adolescents.

ELIGIBILITY:
<Inclusion Criteria>

* Newly diagnosed pediatric/adolescent acute lymphomblastic leukemia patient with NCL standard risk that stratifies all 1-4 of following

  1. 1 year old ≤ Age < 10 years old
  2. white blood cell at initial diagnosis < 5x10^10/L (50,000uL)
  3. No testis involvement
  4. Satisfaction of following organ functions

A. Kidney function (satisfies i or ii) i. Creatinine clearance (or radioisotope-measured GFR) ≥ 70mL/min/1.73m2 ii. Creatinine value according to age/sec satisfies the following:

1 to < 2 years: Male: 0.6 / Female: 0.6, 2 to < 6 years: Male: 0.8 / Female: 0.8, 6 to < 10 years: Male: 1 / Female: 1, 10 to < 13 years: Male: 1.2 / Female: 1.2, 13 to < 16 years: Male: 1.5 / Female: 1.4, ≥ 16 years: Male: 1.7 / Female: 1.4 However, subjects who meet the selection criteria within 1 week before registration after receiving appropriate conservative treatment, including fluid therapy, can be registered.

B. Liver function i. Direct bilirubin < 3.0mg/dL

<Exclusion Criteria>

1. Steroid administration within 2 weeks before the registration
2. t(9;22) or t(4;11)(q11;q23) or chromosome < 44 or iAMP21 or t(17;19)/TCF3-HLF
3. Newly diagnosed T cell ALL
4. One of the following syndromes: Down syndrome, Bloom syndrome, ataxia-telangiectasia, Fanconi anemia, Kostmann syndrome, Shwachman-Diamond syndrome, or other bone marrow failure syndrome
5. Burkitt leukemia/lymphoma
6. In the presence of electrocardiographic findings suggesting uncontrolled cardiac dysfunction (e.g., unstable ischemia, symptomatic arrhythmia, congestive heart failure) or congenital long QT syndrome
7. When the clinical trial subject(or legal representative) does not consent or is unable to give written consent

Ages: 1 Year to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2024-03-05 (Actual); Primary Completion 2033-12-31 (Estimated); Study Completion 2033-12-31 (Estimated)

PRIMARY OUTCOMES:
5-year event free survival rate | Up to 5-years

SECONDARY OUTCOMES:
Confirmation of the therapeutic effect of the initial treatment response | Up to 5-years
  Relapse-free survival between two groups(NGS-MRD positive vs. NGS MRD negative after induction) offsets by NGS MRD based stratified treatment
Disease prognosis-related factor | Up to 5-years
  Relapse-free survival according to presence or absence of known good prognosis factors(high hyperdilpoidy, ETV6/RUNX1, Trisomy 4/10/17) have no clinical significance when NGS MRD based stratified treatment is performed.

CONTACTS AND LOCATIONS:
Locations (9):
- South Korea (9):
  - Asan Medical Center, Seoul, Other (Non U.s.)
  - Samsung Medical Center, Seoul, Other (Non U.s.)
  - Pusan National University Yangsan Hospital, Yangsan, Yangsan-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - Jeju National University Hospital, Jeju City
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Seoul
  - Seoul saint Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided